CLINICAL TRIAL: NCT06259097
Title: Misoprostol Versus Pitocin for Induction of Labor in Patients With BMI > 30: A Randomized Controlled Trial
Brief Title: Different Medications to Induce Labor
Acronym: BLOOM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Bronx Care Health System (Other)
Responsible Party: Principal Investigator, Angela Bianco, Division Director, MFM, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-00118
Record Dates: First submitted 2024-01-29; First posted 2024-02-14 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy; Labor
MeSH Terms: interventions — Misoprostol; Soy Foods; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Misoprostol and Pitocin (Active Comparator): Patient receives misoprostol and foley catheter for initial induction of labor, followed by pitocin later on.
  Interventions: Drug: Misoprostol; Drug: Pitocin
- Pitocin only (Active Comparator): Patient receives pitocin and foley catheter for initial induction of labor, followed by more pitocin later on.
  Interventions: Drug: Pitocin

INTERVENTIONS:
Drug: Misoprostol — 25 mcg vaginally every 6 hours
  Other Names: Miso
  Arms: Misoprostol and Pitocin
Drug: Pitocin — 3-6 mL intravenously every hour

SUMMARY:
This is a randomized controlled trial examining whether the use of misoprostol or pitocin, in combination with a foley catheter, is more effective at inducing labor in patients with a gravid BMI that is considered obese.

DETAILED DESCRIPTION:
This randomized controlled trial will include patients with a BMI greater than 30 at the time of admission for their induction of labor. Patients will be randomized to either misoprostol or Pitocin to begin induction of labor, alongside the standard foley catheter, and the primary outcome of interest will be length of time from start of induction until delivery.

ELIGIBILITY:
Inclusion Criteria:

- Pregnant patient presenting to labor & delivery for induction of labor with a BMI > = 30

Exclusion Criteria:

- Pregnant patient presenting to labor & delivery for induction of labor with BMI < 30

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Time from induction to delivery | start of induction until delivery
  Simple measure calculating time from start of induction until delivery of neonate.

SECONDARY OUTCOMES:
Delivery outcome | at delivery
  Simple determination whether patient had a vaginal delivery or delivered by cesarean section.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola F Tavella, MPH, Study Director — Icahn School of Medicine at Mount Sinai; Angela Bianco, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai Hospital, New York, New York
  - Bronx Care Health System, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  To achieve aims in the approved proposal. Proposals should be directed to Nicola.tavella@mssm.edu. To gain access, data requestors will need to sign a data access agreement.